CLINICAL TRIAL: NCT07029724
Title: Comparison of Standard CPR and CPR Feedback Devices in Terms of the Effectiveness of Chest Compressions During Cardiopulmonary Resuscitation
Brief Title: Effectiveness of Chest Compressions With Standard vs Feedback-Assisted CPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Betül Akbuğa Özel (Other)
Collaborators: Baskent University (Other)
Responsible Party: Sponsor-Investigator, Betül Akbuğa Özel, Assistant Professor, MD, FTBEM, MSc, PhD, Ankara City Hospital Bilkent
Organization: Ankara City Hospital Bilkent (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KA16/73
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: CPR Quality Assessment
Keywords: CPR quality; clinical training; emergency medicine; feedback device; simulation

STUDY DESIGN:
Intervention Model Description: Our study is a randomized trial comparing standard CPR, metronome-guided CPR, and feedback device-assisted CPR (TrueCPR) to enhance the effectiveness of CPR in emergency medicine clinical skills training. It was designed as a single-center, parallel-group, open-label randomized trial. The study design and participant flow diagram were structured in accordance with the CONSORT 2010 guidelines.
Masking Description: Blinding was maintained during data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Standard-to-Metronome Group (Experimental): The Standard-to-Metronome group (Group 1, n = 43) did not have device-specific training and multisensory feedback. In our study, the metronome function was used as a coaching device, optionally integrated with an advanced manikin. This group performed chest compressions without feedback on an advanced manikin, followed by compressions assisted by a metronome providing auditory feedback only, without receiving any device-specific training or multisensory input.
  Interventions: Device: Ambu Smartman ALS Pro+ (AW301) Simulation Manikin; Device: Metronome
- Group 2: Standard-to-TrueCPR Group (Experimental): The Standard-to-TrueCPR Group (Group 2, n = 39) had TrueCPR-specific training and multisensory feedback. TrueCPR is a CPR feedback device equipped with auditory, visual, and cognitive feedback features. Feedback devices monitor each compression and offer corrective information based on real-time performance. This group performed chest-compressions-only CPR without feedback on an advanced manikin, then received training on TrueCPR, and then performed compressions assisted by TrueCPR.
  Interventions: Device: TrueCPR Multisensory Feedback Device; Device: Ambu Smartman ALS Pro+ (AW301) Simulation Manikin

INTERVENTIONS:
Device: TrueCPR Multisensory Feedback Device — TrueCPR (Physio-Control, Inc., Redmond, WA, USA) is a real-time CPR feedback device that provides both visual and auditory cues to support the delivery of high-quality chest compressions. The system consists of two pads (chest and back) that measure compression depth using electromagnetic signal transmission. The device offers auditory rate guidance via a metronome and visual feedback through a color display indicating the adequacy of compression depth and recoil. Performance data-including compression depth, rate, ratio, and the percentage of compressions that are too shallow or too deep-are recorded and analyzed using dedicated software. TrueCPR delivers multisensory feedback (auditory and visual) for both professional rescuers and trainees.
  Arms: Group 2: Standard-to-TrueCPR Group
Device: Ambu Smartman ALS Pro+ (AW301) Simulation Manikin — The Ambu SmartMan ALS Pro+ (AW301) is an advanced simulation manikin designed to support training in both Basic and Advanced Life Support (BLS and ACLS). It features multiple operational modes, including feedback, skills, code, and application modules, with or without manikin dependency. The manikin provides real-time auditory feedback through an integrated metronome and allows online monitoring by instructors. It records performance metrics such as compression depth and rate, compression-to-decompression ratio, hand position accuracy, and number of compressions with leaning.
Device: Metronome — The Ambu SmartMan ALS Pro+ (AW301), which is an advanced simulation manikin, offers real-time auditory feedback via an integrated metronome function. Devices that provide only a fixed auditory tempo-such as a metronome-are generally classified as coaching devices, because they do not measure or analyze the user's actions during CPR.
  Arms: Group 1: Standard-to-Metronome Group

SUMMARY:
The objective of this educational clinical trial is to compare auditory (metronome) and audiovisual (TrueCPR) feedback systems with both standard CPR and with each other in a simulated environment, focusing on their effects on chest compression quality.

The main research questions are:

* Does the use of a metronome improve CPR performance metrics compared to standard CPR?
* Does the use of TrueCPR improve CPR performance metrics compared to standard CPR?
* Is TrueCPR more effective than the metronome in improving CPR performance metrics?

Researchers will evaluate the impact of auditory (metronome) and audiovisual (TrueCPR) feedback systems on chest compression quality by comparing them to standard CPR and to each other within a simulated clinical educational environment.

Participants:

A total of 179 participants, consisting of medical students (n = 112) and paramedic students (n = 67), will be involved in the study.

All participants will attend a 30-minute orientation session. Participants who meet the inclusion criteria and agree to participate (medicine, n = 21; paramedic, n = 62) will sign an informed consent form prior to the study.

They will then complete a preliminary assessment, including a 5-question knowledge test on high-quality CPR metrics.

Perform 2 minutes of chest-compressions-only CPR (standard CPR) on a manikin without any feedback.

All participants will be pooled and randomized. They will receive a 10-minute general briefing session after randomization.

Study Groups:

Group1: Standard-to-Metronome Group (n = 43) will:

Perform 2 minutes of chest-compressions-only CPR (standard CPR) on a manikin without any feedback.

Not receive device-specific training or use a multisensory feedback device. Take a 5-minute rest period. Perform 2 minutes of CPR using metronome feedback.

Group 2: Standard-to-TrueCPR (n = 40) will:

Perform 2 minutes of chest-compressions-only CPR (standard CPR) on a manikin without any feedback.

Receive a 30-minute TrueCPR-specific training session and use a multisensory feedback device.

Take a 5-minute rest period. Perform 2 minutes of CPR using TrueCPR feedback.

DETAILED DESCRIPTION:
A. Study Preparation Study Setting This study was conducted in the Professional Skills Laboratories of Başkent University Faculty of Medicine. Basic Life Support (BLS) simulations were organized as standardized, single-station sessions and performed on an advanced ACLS manikin situated in a spacious hands-on training room. While one participant performed chest compressions, others waited in a nearby area until it was their turn.

Research Personnel Two faculty members designed the simulation environment and BLS scenarios, supervised orientation training for both investigators and participants, and coordinated study sessions. Additionally, five medical student researchers assisted in setting up the simulation environment, managing participant flow, delivering orientation sessions, and obtaining informed consent.

Orientation Session A 30-minute orientation session was held on two separate days for the study population (medicine, n = 112; paramedic, n = 67), during which the study purpose, pre- and post-randomization procedures, study setting, and participant expectations were explained.

Preliminary Assessment Before the randomization phase, a preliminary assessment was conducted to evaluate the similarities in high-quality CPR knowledge and performance between medical and paramedic students.

* Participants who attended the orientation were invited to participate in the study (n = 83). Demographic data were collected, and informed consent was obtained from volunteers meeting the inclusion criteria (medicine, n = 21; paramedic, n = 62).
* A five-question knowledge test covering key high-quality CPR metrics was administered. The test scores were recorded for all eligible participants.
* Each participant then performed 2 minutes of chest-compressions-only CPR on an advanced ACLS manikin without feedback. Compression rate, depth, and residual leaning percent were recorded for each participant.
* Knowledge test and performance data were analyzed separately for medical and paramedic students.
* Analyses showed no significant differences in theoretical knowledge or practical performance between the two groups.
* Due to this equivalence, participants were pooled and randomized irrespective of their educational background.

Randomization

Two sets of labels were prepared: one labeled "standard to metronome" and "standard to TrueCPR," and the other labeled "Group 1" and "Group 2." These were matched by blind draw to assign the intervention types to each group:

Group 1: Metronome group, "Standard to Metronome" (no device-specific training or multisensory feedback) Group 2: TrueCPR group, "Standard to TrueCPR" (device-specific training and audiovisual feedback)

Of 179 eligible participants, 83 met the inclusion criteria, demonstrated equivalent knowledge and performance, gave informed consent, and were randomized. A block randomization method (1:1 ratio) was implemented using a web-based tool (Urbaniak GC, http://www.randomizer.org/) to ensure balanced allocation. Participants were assigned to either Group 1 (n = 43) or Group 2 (n = 40). The slight imbalance reflected differences in enrollment timing and participant availability and was acceptable within block design limits.

To maintain allocation concealment, the randomization sequence was generated and managed by an independent researcher not involved in recruitment or data collection. The allocation list was stored securely and remained inaccessible to investigators until the assignment.

Because standard CPR, metronome-assisted CPR, and TrueCPR-assisted CPR are clearly distinguishable in cognitive, visual, and auditory dimensions, the study was conducted as open-label for researchers, participants, and the data analyst.

B. Study Interventions Group assignments were performed by an independent researcher prior to the start of the trial to ensure unbiased allocation.

Group 1 (n = 43): Performed chest-compressions-only CPR (standard CPR) followed by metronome-assisted CPR, without receiving any specific training or multisensory feedback.

Group 2 (n = 40): Performed device-specific training (TrueCPR) and performed chest-compressions-only CPR (standard CPR) followed by TrueCPR-assisted CPR with auditory and visual feedback. In this group, one participant did not complete the CPR session with TrueCPR.The number of participants included in the analyses was 39 (n = 39).

Intervention Steps

1. At the beginning of the trial, both groups received a standardized 10-minute briefing, including an overview of the study protocol, orientation to the simulation lab, and introduction to the research team.
2. In a single-station setup:

   Group 1 participants first performed 2 minutes of standard CPR without ventilation or feedback. After a 5-minute rest, they performed another 2 minutes of CPR assisted by a metronome. The metronome feature was embedded in the advanced ACLS manikin and provided auditory feedback only. No additional training was given.
3. On a different day, using the same station:

   Group 2 participants first performed 2 minutes of standard CPR without feedback. Then, they received a 30-minute device-specific TrueCPR training, which included:

   A 10-minute instructional video, A 10-minute didactic session, A 5-minute demonstration and Q&A session, A 2-minute individual hands-on practice, A 5-minute rest period. Finally, they performed 2 minutes of CPR using the TrueCPR device, which provided real-time audiovisual feedback.
4. Chest compression rate (cpm), depth (mm), and leaning percent (%) were measured and recorded during standard CPR, metronome-guided CPR, and TrueCPR-assisted CPR using the Ambu SmartMan ALS Pro+ (AW301) manikin.

ELIGIBILITY:
Inclusion Criteria:

* Being a first- or second-year student in the medical school or paramedic program
* Having completed a standardized Basic Life Support (BLS) course as part of the curriculum
* Having no prior experience with CPR feedback devices
* Voluntarily agreeing to participate and signing the informed consent form
* Being able to complete all required chest compression steps during the study procedure

Exclusion Criteria:

* Being a student other than first- or second-year in the medical school or paramedic program
* Not having completed a standardized Basic Life Support (BLS) course as part of the academic curriculum
* Having prior experience with CPR feedback devices
* Refusing to participate or failing to sign the informed consent form
* Being unable to perform all required chest compression steps during the study procedure

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-04-22 (Actual); Primary Completion 2016-05-02 (Actual); Study Completion 2016-05-02 (Actual)

PRIMARY OUTCOMES:
Chest compression rate | From randomization to the completion of all chest compression procedures, within a maximum duration of 60 minutes.
  One of the primary outcomes of the study was the chest compression (CC) rate, measured in compressions per minute (cpm). According to the 2020 American Heart Association (AHA) Guidelines for Cardiopulmonary Resuscitation, a key component of high-quality CPR is maintaining an optimal CC rate of 100 to 120 cpm in adult patients. This rate ensures sufficient blood flow during cardiac arrest while minimizing the risk of inadequate ventricular filling. In our study, CC rate outcomes were objectively measured and recorded using the Ambu SmartMan ALS Pro+ (AW301) manikin.
Chest compression depth | From randomization to the completion of all chest compression procedures, within a maximum duration of 60 minutes.
  One of the primary outcomes of the study was the chest compression (CC) depth, measured in millimeters (mm). According to the 2020 American Heart Association (AHA) Guidelines, high-quality CPR requires a CC depth of 5 to 6 centimeters (50-60 millimeters) in adults to ensure adequate blood flow during resuscitation. In this study, CC depth outcomes were measured and recorded using the Ambu SmartMan ALS Pro+ (AW301) manikin.
Leaning percent | From randomization until the end of the chest compression sessions, within a 60-minute period.
  One of the primary outcomes of the study was the Leaning Percent (LP), measured as a percentage (%). According to the 2020 American Heart Association (AHA) Guidelines for Cardiopulmonary Resuscitation, complete release after each compression is essential to ensure optimal cardiac filling and perfusion. Leaning percent reflects how often chest compressions are performed without allowing full chest recoil. Incomplete release can compromise the effectiveness of CPR. In this study, the Ambu SmartMan ALS Pro+ (AW301) manikin automatically recorded the number of compressions with incomplete release during each 120-second chest-compression-only session. The LP was calculated using the formula: Leaning % = (Compressions with incomplete release / Total compressions) × 100.

CONTACTS AND LOCATIONS:
Overall Officials: Betül Akbuğa Özel, Asst. Prof., Principal Investigator — Ankara Yıldırım Beyazıt University, Faculty of Medicine, Ankara Bilkent City Hospital, Department of Emergency Medicine
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Bilkent City Hospital, Ankara Yıldırım Beyazıt University, Faculty of Medicine, of Emergency Medicine, Çankaya, Ankara
  - Başkent University, Etimesgut, Ankara

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to share individual participant data (IPD). As the data are the property of Başkent University, any decision regarding access must be made at the institutional level. During the publication process of the study, IPD may be shared upon request to the principal investigator and is subject to institutional approval.

REFERENCES:
- [Background] Smereka J, Szarpak L, Czekajlo M, Abelson A, Zwolinski P, Plusa T, Dunder D, Dabrowski M, Wiesniewska Z, Robak O, Frass M, Sivrikaya G U, Ruetzler K. The TrueCPR device in the process of teaching cardiopulmonary resuscitation: A randomized simulation trial. Medicine (Baltimore). 2019 Jul;98(27):e15995. doi: 10.1097/MD.0000000000015995. PMID 31277091
- [Background] Lin Y, Lockey A, Donoghue A, Greif R, Cortegiani A, Farquharson B, Siddiqui FJ, Banerjee A, Matsuyama T, Cheng A; Education Implementation Team Task Force of the International Liaison Committee on Resuscitation ILCOR. Use of CPR feedback devices in resuscitation training: A systematic review and meta-analysis of randomized controlled trials. Resusc Plus. 2025 Mar 22;23:100939. doi: 10.1016/j.resplu.2025.100939. eCollection 2025 May. PMID 40230367
- [Background] Zapletal B, Greif R, Stumpf D, Nierscher FJ, Frantal S, Haugk M, Ruetzler K, Schlimp C, Fischer H. Comparing three CPR feedback devices and standard BLS in a single rescuer scenario: a randomised simulation study. Resuscitation. 2014 Apr;85(4):560-6. doi: 10.1016/j.resuscitation.2013.10.028. Epub 2013 Nov 8. PMID 24215730
- [Background] Szarpak L, Bogdanski L, Czyzewski L, Zasko P, Kurowski A. Are chest compressions using the TrueCPR feedback device more effective than manual compressions during pediatric resuscitation? A randomized controlled trial. Indian Journal of Research. 2015; 4(1):84-86.
- [Background] Wutzler A, Bannehr M, von Ulmenstein S, Loehr L, Forster J, Kuhnle Y, Finn A, Storm C, Haverkamp W. Performance of chest compressions with the use of a new audio-visual feedback device: a randomized manikin study in health care professionals. Resuscitation. 2015 Feb;87:81-5. doi: 10.1016/j.resuscitation.2014.10.004. Epub 2014 Oct 17. PMID 25449342
- [Background] Kurowski A, Szarpak L, Bogdanski L, Zasko P, Czyzewski L. Comparison of the effectiveness of cardiopulmonary resuscitation with standard manual chest compressions and the use of TrueCPR and PocketCPR feedback devices. Kardiol Pol. 2015;73(10):924-30. doi: 10.5603/KP.a2015.0084. Epub 2015 May 19. PMID 25985725
- [Background] Truszewski Z, Szarpak L, Kurowski A, Evrin T, Zasko P, Bogdanski L, Czyzewski L. Randomized trial of the chest compressions effectiveness comparing 3 feedback CPR devices and standard basic life support by nurses. Am J Emerg Med. 2016 Mar;34(3):381-5. doi: 10.1016/j.ajem.2015.11.003. Epub 2015 Nov 4. PMID 26612703
- [Background] Panchal AR, Bartos JA, Cabanas JG, Donnino MW, Drennan IR, Hirsch KG, Kudenchuk PJ, Kurz MC, Lavonas EJ, Morley PT, O'Neil BJ, Peberdy MA, Rittenberger JC, Rodriguez AJ, Sawyer KN, Berg KM; Adult Basic and Advanced Life Support Writing Group. Part 3: Adult Basic and Advanced Life Support: 2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2020 Oct 20;142(16_suppl_2):S366-S468. doi: 10.1161/CIR.0000000000000916. Epub 2020 Oct 21. No abstract available. PMID 33081529
- See also: Smereka J, Szarpak L, Czekajlo M, Abelson A, Zwolinski P, Plusa T, et al. The TrueCPR device in the process of teaching cardiopulmonary resuscitation: A randomized simulation trial. Medicine (Baltimore). 2019 Jul;98(27):e15995. — https://pmc.ncbi.nlm.nih.gov/articles/PMC6635263/pdf/medi-98-e15995.pdf